CLINICAL TRIAL: NCT06683469
Title: Neutrophil-to-Lymphocyte Ratio in Predicting Outcomes of Patients With Aneurysmal Subarachnoid Hemorrhage in a Tertiary Care Hospital in Nepal
Status: Completed | Type: Observational
Sponsor: Sujan Paudel (Other)
Responsible Party: Sponsor-Investigator, Sujan Paudel, Dr, Maharajgunj Medical Campus
Organization: Maharajgunj Medical Campus (Other)
Other Study IDs: MaharajgunjMed
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: SAH (Subarachnoid Hemorrhage)
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study uses Neutrophil-to-Lymphocyte Ratio to Predict Outcomes of Patients with Aneurysmal Subarachnoid Hemorrhage which will be beneficial in taking early decisions for surgery , patient counselling etc

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age, of either genders, ethnicity and location who presented to the emergency department within 72 hours of the onset of symptoms who underwent surgical or interventional treatment for SAH caused by a ruptured intracranial aneurysm

Exclusion Criteria:

* excluded patients with traumatic SAH, history of infection or stroke within eight weeks, underlying cancer, severe kidney or liver disease, history of auto-immune or hematologic disorder lost to follow-up within three months and individuals declining informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years of age, of either genders, ethnicity and location who presented to the emergency department within 72 hours of the onset of symptoms who underwent surgical or interventional treatment for SAH caused by a ruptured intracranial aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
mRS score | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Guo Y, Liu J, Zeng H, Cai L, Wang T, Wu X, Yu K, Zheng Y, Chen H, Peng Y, Yu X, Yan F, Cao S, Chen G. Neutrophil to lymphocyte ratio predicting poor outcome after aneurysmal subarachnoid hemorrhage: A retrospective study and updated meta-analysis. Front Immunol. 2022 Aug 9;13:962760. doi: 10.3389/fimmu.2022.962760. eCollection 2022. PMID 36016932